CLINICAL TRIAL: NCT00962468
Title: The European Quality of Care Pathways Study: The Impact of a Care Pathway for Exacerbation of Chronic Obstructive Pulmonary Disease (COPD) : an International Cluster Randomized Controlled Trial." (Www.E-P-A.Org)
Brief Title: European Quality of Care Pathways Study on Chronic Obstructive Pulmonary Disease (COPD)
Acronym: EQCP-COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Pathway Association (Other)
Collaborators: KU Leuven (Other); University of Eastern Piedmont (Other)
Responsible Party: Principal Investigator, Dr. Kris Vanhaecht, Dr. Kris Vanhaecht, Secretary General, European Pathway Association, ivzw, European Pathway Association
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EPA-EQCP001
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Critical Pathway; Cluster Randomized Controlled Trial; Safety; Efficiency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Critical Pathways

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pathway (Experimental): A care pathway will be implemented in this experimental group.
  Interventions: Other: COPD evidence based care pathway
- Usual care (No Intervention): Usual care will be provided.

INTERVENTIONS:
Other: COPD evidence based care pathway — A care pathways, as complex intervention, will be implemented.
  Other Names: pathway; care pathway; clinical pathway; critical pathway; integrated care pathway
  Arms: Pathway

SUMMARY:
Care pathways, a complex intervention to (re)organise, standardize and evaluate care processes, are used worldwide and in different kinds of settings. Although their international use, the impact is unclear. The European Quality of Care Pathways Study is the first international cluster Randomized Controlled Trial on the effect of care pathways for COPD patients.

The hypothesis is that teams who work with care pathways for COPD patients deliver care that is more compliant to evidence based key interventions, have better patient outcomes and higher scores on team indicators than teams who do not work with care pathways.

DETAILED DESCRIPTION:
Healthcare is changing towards more patient focused care. The organization of the care process related to quality, efficiency and accessibility is one of the main areas of interest within the next years for clinicians, healthcare managers and policy makers. A main method to (re)organize a care process is the development and implementation of a care pathway. Care pathways, also known as clinical pathways or critical pathways, are used worldwide for a variety of patient groups. The European Pathway Association (E-P-A) defines a care pathway as: "A complex intervention for the mutual decision making and organization of predictable care for a well-defined group of patients during a well defined period. Defining characteristics of pathways includes: an explicit statement of the goals and key elements of care based on evidence, best practice and patient expectations; the facilitations of the communication and coordination of roles, and sequencing the activities of the multidisciplinary care team, patients and their relatives; the documentation, monitoring, and evaluation of variances and outcomes; and the identification of relevant resources".

Very few prospective studies have been performed and published on the impact of pathways on quality and efficiency of care. The European Quality of Care Pathways (EQCP)-study will involve exacerbation of Chronic Obstructive Pulmonary Disease (COPD) to evaluate pathway effectiveness. Literature shows that adherence to international guidelines with regard to inhospital management of COPD exacerbation is low, especially in non pharmacological treatment.11-19 Currently, only three non-randomized trials about the impact of a care pathway for inpatient management of COPD exacerbation are published. The studies are conducted between 1995 and 2001, and the methodology is doubtful. However the studies indicate that a COPD exacerbation care pathway improves performance with regard to diagnostic assessment and use of standing orders, and that it diminishes the number of rehospitalisation, shortens length of stay (LOS) and reduces mortality.

In the context of the high volume of hospitalized COPD patients, high costs and high risk, and the complex coordination of care among multiple caregivers, a care pathway could enhance the quality of care in these patients by improving patient outcomes, promoting patient safety, increasing patient satisfaction, improving multidisciplinary teamwork and optimizing the use of resources.

The goal of the European Quality of Care Pathways (EQCP) study is:

* To evaluate the care pathway effectiveness in acute hospitals and their immediate link with primary care;
* To evaluate the effect of care pathways on team processes and team perceived organization of care.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria on cluster level are:

1. Written agreement to participate in the study;
2. Agreement that a care pathway for COPD will not be developed and used within the time frame of the study when randomized in the control group.

Inclusion criteria on patient level are:

1. Written informed consent;
2. All consecutive admissions with COPD exacerbation;
3. Hospitalization for at least 48 hours;
4. Moderate, severe or very severe COPD;
5. Each patient will be included only once in the study at initial hospitalization, even if the patient had been hospitalized more than once.

Exclusion Criteria:

Exclusion criteria on patient level:

1. Admission required to intensive care unit;
2. Need for Invasive Positive Pressure Ventilation (IPVV).

Inclusion criteria on multidisciplinary team level:

1. Team members are involved in direct patient care responsibilities for COPD;
2. Minimum representation of the core disciplines according to COPD literature;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2009-05; Primary Completion 2014-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Readmission rate | 6 month

SECONDARY OUTCOMES:
Mortality | 1 year
Length of stay | in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Kris Vanhaecht, PhD, Study Director — KU Leuven; Walter Sermeus, PhD, Principal Investigator — KU Leuven; Massimiliano Panella, PhD, Principal Investigator — Amedeo Avogadro University of Eastern Piemont

REFERENCES:
- [Derived] Vanhaecht K, Sermeus W, Peers J, Lodewijckx C, Deneckere S, Leigheb F, Decramer M, Panella M; EQCP Study Group. The impact of care pathways for exacerbation of Chronic Obstructive Pulmonary Disease: rationale and design of a cluster randomized controlled trial. Trials. 2010 Nov 19;11:111. doi: 10.1186/1745-6215-11-111. PMID 21092098
- See also: European Pathway Association — http://www.E-P-A.org